CLINICAL TRIAL: NCT06928181
Title: Effects of Passive Blood-Flow-Restriction Training on Muscle Atrophy and Pain After Elective Total Knee Arthroplasty
Brief Title: Effects of Passive Blood-Flow-Restriction on Muscle Atrophy and Pain After Elective Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023_A_TKA_BFR
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis in the Knee
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Sham-BFR Intervention with 20mmHg
  Interventions: Other: Sham-BFR
- Intervention (Experimental): BFR-Intervention with 80% of the 1RM
  Interventions: Other: Blood Flow Restriction Training

INTERVENTIONS:
Other: Blood Flow Restriction Training — BFR training involves the application of blood flow restriction during passive or active movement interventions to elicit an additional metabolic stimulus. The cuffs are applied as proximally as possible on the thigh, and a pressure is exerted during the movement that partially restricts venous return from the limb, resulting in venous pooling. Venous occlusion is achieved using a cuff system commonly employed in resistance training (Delfi Medical Innovations Inc., Vancouver, Canada; CE-certified). The pressure applied is individually determined at the start of each training session based on the participant's arterial occlusion pressure, measured via duplex ultrasonography. For this measurement, the participant rests in a supine position while the cuff is gradually inflated until no blood flow is detectable in the limb (i.e., occlusion pressure). For the BFR intervention, 60-80% of this occlusion pressure is subsequently applied. The exercise protocol consists of daily
  Arms: Intervention
Other: Sham-BFR — Patients in the control group (CG) follow the same exercise protocol as those in the BFR intervention group; however, the cuff is only inflated to a minimal pressure of 20 mmHg. This pressure does not induce any relevant venous stasis, nor can any local or systemic metabolic effects be expected.
  Arms: Control

SUMMARY:
This study investigated the effects of passive Blood-Flow-Restriction Training after elective Total Knee Arthroplasty Surgery on Muscle Atrophy and Postoperative Pain.

DETAILED DESCRIPTION:
This is the first study invesigating the effects of passive Blood-Flow-Restriction Training on Muscle Atrophy and Postoperative Pain after Elective Total Knee Arthroplasty Surgery.

ELIGIBILITY:
Inclusion Criteria:

* The study includes all patients with a medical indication for surgical treatment of the lower extremity (total or partial knee arthroplasty) who are eligible for either inpatient or outpatient rehabilitation.
* All participating patients have signed the informed consent form for study participation as well as the data protection declaration after receiving comprehensive explanation, counseling, and information.
* All patients have consented to the surgical procedure and received medical clearance for surgery from both the orthopedic and anesthesiology departments.

Exclusion Criteria:

* Acute or chronic infections of the extremities
* Open wounds on the lower extremity
* Pregnancy and breastfeeding
* Patients who are unable to understand the patient information and study design (e.g., due to language barriers), or whose compliance is deemed insufficient by the study team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Muscle Mass | Three Months
  Lean Body Mass in DEXA anaylsis
Postoperative Pain | Three Months
  0-100 mm VAS

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No